CLINICAL TRIAL: NCT00900406
Title: Tissue Bank for Studies Related to Graft-Versus-Host Disease (GVHD)
Brief Title: Collecting and Storing Tissue and DNA Samples From Patients Undergoing a Donor Stem Cell Transplant
Status: Completed | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Madan Jagasia, MD, Associate Professor of Medicine; Director, Outpatient Transplant Program; Section Chief, Hematology and Stem Cell Transplant;, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC BMT 0664; P30CA068485 (NIH); VU-VICC-BMT-0664; VU-VICC-IRB-061215
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Breast Cancer; Chronic Myeloproliferative Disorders; Gestational Trophoblastic Tumor; Graft Versus Host Disease; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; Neuroblastoma; Ovarian Cancer; Testicular Germ Cell Tumor
MeSH Terms: conditions — Breast Neoplasms; Myeloproliferative Disorders; Gestational Trophoblastic Disease; Graft vs Host Disease; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Neuroblastoma; Ovarian Neoplasms; Testicular Germ Cell Tumor | interventions — Gene Expression Profiling; Microarray Analysis; Amplified Fragment Length Polymorphism Analysis; Flow Cytometry; Immunologic Techniques; Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood collection

GROUPS / COHORTS (3):
- Recipients of stem cells with graft versus host disease
  Interventions: Genetic: gene expression analysis; Genetic: microarray analysis; Genetic: polymorphism analysis; Genetic: proteomic profiling; Other: flow cytometry; Other: immunologic technique; Other: laboratory biomarker analysis; Procedure: biopsy
- Recipients of stem cells at risk of graft versus host disease
  Interventions: Genetic: gene expression analysis; Genetic: microarray analysis; Genetic: polymorphism analysis; Genetic: proteomic profiling; Other: flow cytometry; Other: immunologic technique; Other: laboratory biomarker analysis; Procedure: biopsy
- Donator of stem cells
  Interventions: Genetic: gene expression analysis; Genetic: microarray analysis; Genetic: polymorphism analysis; Genetic: proteomic profiling; Other: flow cytometry; Other: immunologic technique; Other: laboratory biomarker analysis; Procedure: biopsy

INTERVENTIONS:
Genetic: gene expression analysis — blood collection
Genetic: microarray analysis — Blood collection
Genetic: polymorphism analysis — Blood collection
Genetic: proteomic profiling — Blood collection
Other: flow cytometry — Blood collection
Other: immunologic technique — Blood collection
Other: laboratory biomarker analysis — Blood collection
Procedure: biopsy — Blood collection

SUMMARY:
RATIONALE: Collecting and storing samples of blood, urine, and tissue from patients undergoing a donor stem cell transplant to test in the laboratory may help the study of graft-versus-host disease in the future.

PURPOSE: This research study is collecting and storing tissue and DNA samples from patients undergoing a donor stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

* To establish a DNA bank from donor and recipient (prior to transplant) peripheral blood for SNP studies.
* To establish a tissue bank for gene expression studies using donor and recipient (post-transplant) peripheral blood samples.
* To establish a tissue bank for proteomic studies using donor and recipient blood and urine samples.
* To establish a tissue bank for various studies using biopsy specimens.
* To establish a tissue bank for flow cytometric studies using recipient (post-transplant), and sample from stem cell product.

OUTLINE: Peripheral blood samples are collected from donors prior to stem cell mobilization and from patients prior to starting preparative regimen. Samples are studied by single nucleotide polymorphism (SNP) analysis, SNP array, proteomic analysis, gene expression, and other immunological laboratory methods. Blood, urine, and tissue samples are preserved for future studies. Extra skin biopsies and gastrointestinal biopsies are performed at diagnosis of graft-vs-host disease and preserved in a tissue bank for flow cytometric studies.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Approved for allogeneic stem cell transplantation
* Sample of the stem cells from donor must meet 1 of the following criteria:

  * Total peripheral blood stem cell dose > 5 X10^6 CD34+ cells/kg
  * Marrow cell dose > 3 X 10^8 nucleated cells/kg

PATIENT CHARACTERISTICS:

* Platelet count > 50,000/mm³ (for patients undergoing endoscopic biopsies)
* INR < 1.5 (for patients undergoing endoscopic biopsies)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who have received a stem cell transplant and are being treated for graft versus host disease or are at risk of graft versus host disease.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2007-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
DNA bank from donor and recipient (prior to transplant) peripheral blood for single nucleotide polymorphism studies | Completion of transplant
Tissue bank for gene expression studies using donor and recipient (post-transplant) peripheral blood samples | End of treatment
Tissue bank for proteomic studies using donor and recipient blood and urine samples | End of treatment
Tissue bank for flow cytometric studies using recipient (post-transplant), and sample from stem cell product | End of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Madan Jagasia, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee